CLINICAL TRIAL: NCT02880982
Title: Trial of Vitamin D Supplementation in Cape Town Primary Schoolchildren
Acronym: ViDiKids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 9408
Record Dates: First submitted 2016-07-18; First posted 2016-08-26 (Estimated); Last update posted 2022-09-08 (Actual); Status verified 2022-01

CONDITIONS: Latent Tuberculosis
MeSH Terms: conditions — Latent Tuberculosis | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Softgel capsule containing 10,000 IU (250 micrograms) cholecalciferol (vitamin D3) to be taken orally once per week for 3 years
  Interventions: Dietary Supplement: Cholecalciferol
- Placebo (Placebo Comparator): Softgel capsule of identical taste and appearance to active comparator, but containing no cholecalciferol, to be taken orally once per week for 3 years
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — Weekly oral softgel capsule containing 10,000 IU (250 micrograms) cholecalciferol (vitamin D3)
  Other Names: Vitamin D3
  Arms: Intervention
Other: Placebo — Weekly oral placebo softgel capsule
  Arms: Placebo

SUMMARY:
The investigators will conduct a n=5,400 Phase 3, double-blind, individually randomised placebo-controlled clinical trial of 5 years' duration in primary schools in City of Cape Town Metropolitan Municipality, Western Cape Province, Republic of South Africa.

The primary objective of the trial is to determine whether a weekly oral dose of 0.25 mg (10,000 IU) vitamin D3, administered for three years, reduces risk of acquisition of latent tuberculosis infection (LTBI) in Cape Town primary schoolchildren.

Statistical analysis will be performed on an intention-to-treat basis to compare acquisition of LTBI in intervention vs. control arms during three-year follow-up. The primary analysis will be logistic regression with presence/absence of LTBI at follow-up as the outcome, adjusted for a random effect of school of attendance.

ELIGIBILITY:
Inclusion Criteria:

* Pupil enrolled in Grades 1-4 of participating primary schools
* Age 6-11 years at enrolment
* Pupil gives written informed assent to participate in main trial
* Pupil's parent / legal guardian gives informed consent for pupil to participate in main trial

Exclusion Criteria:

* Age ≤5 years or ≥12 years at enrolment
* Previous positive Interferon-Gamma Release Assay (IGRA) or Mantoux test
* Previous treatment for LTBI or active TB
* Clinical signs of rickets
* History of myalgia on walking
* Inability to rise unaided from squatting position
* Taking supplemental vitamin D at a dose >400 IU daily or equivalent in the previous month
* Diagnosis of any chronic illness other than asthma
* Suspected HIV infection in child with parent or legal guardian declining to have child HIV-tested
* Use of any regular medication other than asthma medication
* Plans to move away from study area within 3 years of enrolment
* Unable to swallow one placebo softgel with ease
* Positive Quantiferon-TB Gold Plus test at screening

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1743 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Acquisition of latent tuberculosis infection | 3 years

SECONDARY OUTCOMES:
Incidence of active tuberculosis (TB) | 3 years
Incidence of acute respiratory infection | 3 years
Incidence of acute asthma exacerbation | 3 years
Incidence and control of asthma, allergic rhinitis and atopic dermatitis | 3 years
Incidence of bone fracture | 3 years
Anthropometric outcomes (weight, height, body mass index, waist circumference) | 3 years
Mathematics examination result | 3 years
Stage of pubertal development, self-assessed using the Tanner scale | 3 years
Bone mineral content, lumbar spine and whole body minus head | 3 years
Body composition including fat mass and fat-free soft tissue mass | 3 years
Muscle strength (grip strength, elastic leg strength) | 3 years
Estimated maximal oxygen uptake, derived from 20 meter shuttle test performance | 3 years
Bronchial hyper-responsiveness to exercise | 3 years
Sensitisation to aeroallergens | 3 years
Concentrations of antigen-stimulated inflammatory mediators | 3 years
Vitamin D status, parathyroid hormone and circulating markers of bone formation and modelling | 3 years
Attention Deficit Hyperactivity Disorder Rating Scale-IV score | 3 years
Cost-effectiveness of vitamin D3 for prevention of LTBI and active TB | 3 years
Incidence of potential adverse reactions to vitamin D3 | 3 years
Incidence of serious adverse events due to any cause | 3 years
Incidence of fatal or life-threatening serious adverse events due to any cause | 3 years
Proportion of participants sero-positive for SARS-CoV-2 at follow-up | 3 years
Proportion of participants sero-positive for seasonal coronaviruses HKU1, 229E, OC43 and NL63 at follow-up | 3 years
Proportion of participants sero-positive for influenza A and B at follow-up | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Keren Middelkoop, MPH, PhD, Principal Investigator — University of Cape Town
Locations (1):
- Desmond Tutu HIV Foundation, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Middelkoop K, Micklesfield L, Stewart J, Walker N, Jolliffe DA, Mendham AE, Coussens AK, Nuttall J, Tang J, Fraser WD, Momand W, Cooper C, Harvey NC, Wilkinson RJ, Bekker LG, Martineau AR. Influence of vitamin D supplementation on growth, body composition, pubertal development and spirometry in South African schoolchildren: a randomised controlled trial (ViDiKids). BMJ Paediatr Open. 2024 Apr 10;8(1):e002495. doi: 10.1136/bmjpo-2024-002495. PMID 38599800